CLINICAL TRIAL: NCT04577729
Title: INDUCING REMISSION IN MELANOMA PATIENTS WITH CHECKPOINT INHIBITOR THERAPY USING FECAL MICROBIOTA TRANSPLANTATION.
Brief Title: The IRMI-FMT Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Agreement with project partner prematurely cancelled.
Sponsor: Medical University of Graz (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA-209-7HP
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Fecal Microbiota Transplantation; Malignant Melanoma Stage III; Malignant Melanoma Stage IV
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Allogenic FMT group (Experimental): Allogenic FMT group: patients receiving stool from prior malignant melanoma (MM) patients in remission for at least 1 year after Checkpoint Inhibitor Treatment.
  Interventions: Procedure: Allogenic Fecal Microbiota Transplantation
- Autologous FMT group (Placebo Comparator): Autologous FMT group: patients receiving their own stool in terms of sham FMT.
  Interventions: Procedure: Autologous Fecal Microbiota Transplantation

INTERVENTIONS:
Procedure: Allogenic Fecal Microbiota Transplantation — Patients receiving stool from prior malignant melanoma (MM) patients in remission for at least 1 year after Checkpoint Inhibitor Treatment.
  Arms: Allogenic FMT group
Procedure: Autologous Fecal Microbiota Transplantation — Patients receiving their own stool in terms of sham FMT.
  Arms: Autologous FMT group

SUMMARY:
Aim of the study is to investigate the effect of Fecal Microbiota Transplantation (FMT) and Checkpoint Inhibitor (CI) re-challenge in prior CI refractory patients on Progression free survival (PFS) and tumor using donor stool of former malignant melanoma patients, who have been in remission due to CI treatment for at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed malignant melanoma

   * Age > 18 years
   * Written consent of the participant after being informed
   * Contraception as described in protocol appendix section VI
2. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS): PS 0 to 1.
3. Previously treated, unresectable stage III or stage IV melanoma as per the American Joint Committee on Cancer 2017 Guidelines (8th Edition) regardless of BRAF mutation status.
4. Patients must have experienced disease progression or recurrence during treatment with an anti-PD-1 monoclonal antibody, not having OR not willing to accept other approved systemic treatment options (like: BRAF and MEK inhibitors in BRAF V600 mutated melanoma).
5. Patients with CNS (central nervous system) metastases:

   * Patients are eligible if CNS metastases are treated and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks Prior to enrolment. In addition, patients must be either off corticosteroids or on a stable or decreasing dose <10 mg daily prednisone (or equivalent) OR
   * Patients are eligible if they have previously untreated CNS metastases and are neurologically asymptomatic. In addition, patients must be either off corticosteroids or on a stable or decreasing dose of <10 mg daily prednisone (or equivalent) OR
   * Patients with additional leptomeningeal metastases are eligible if they are treated and neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment) for at least 2 weeks prior to enrolment and have an estimated life expectancy of at least 3 months. In addition, subjects must be either off corticosteroids or on a stable or decreasing dose of <10 mg daily prednisone (or equivalent)
6. Patients must have evaluable disease by CT (computer tomography) or MRI (magnet resonance imaging) per RECIST 1.1 criteria (Appendix 3) (radiographic tumor assessment performed before as well as after 10 weeks of first dose of study drug) or clinically apparent disease that the investigator can follow for response.

Exclusion Criteria:

1. Active brain metastases or leptomeningeal metastases. Participants with brain metastases are eligible if these have been treated and there is no MRI evidence of progression for at least 2 weeks after treatment is complete and within 28 days prior to first dose of study treatment administration. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (> 10 mg/day prednisone equivalents) for at least 2 weeks prior to study treatment administration. Stable dose of anticonvulsants is allowed. Treatment for CNS metastases may include stereotactic radiosurgery (e.g. GammaKnife, CyberKnife, or equivalent) or neurosurgical resection. Patients who received whole brain radiation therapy are not eligible.
2. Prior treatment with chemotherapy, interferon (adjuvant setting), IL-2 (Interleukin-2), BRAF/MEK Inhibitors (v-Raf murine sarcoma viral oncogene homolog B/Mitogen-Activated Protein Kinase) for subjects with known BRAF V600 mutations, MEK inhibitors for NRAS (N-Rat sarcoma) mutations, and cKIT (Tyrosinkinase) Inhibitor subjects with known cKIT mutations is NOT allowed.
3. Uveal melanoma is excluded.
4. Coexisting severe chronic diseases other than melanoma (other neoplasias, autoimmune diseases,…).
5. Secondary gastrointestinal motility disorders.
6. Pregnancy and breast feeding.
7. Large abdominal surgery in medical history.
8. Intake of any medication introduced by another clinical study.
9. Any conditions (e.g. allergies), that do not allow the administration or intake of any of the substances used in this study (Nivolumab, Vancomycin, colonic lavage fluid).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-06-07 (Actual); Study Completion 2023-06-07 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 3 months after checkpoint inhibitor (CI) therapy following fecal microbiota transplantation (FMT).
  Patients undergoing CI therapy after FMT will be evaluated by Immune-RECIST (iRECIST) criteria after contrast-enhanced CT-scan in order to determine disease progression.

SECONDARY OUTCOMES:
Tumor response (CR, PR, SD) | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  Complete response (CR), partial response (PR) and stable disease (SD) of target or non-target lesions are considered tumor response in this trial according to iRECIST criteria after three months.
Detection of specific donor signaling in intestinal microbiota leading to response to CI therapy. | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  A total of five donors will be included in the study. The allogenic-FMT group will receive donor stool from a single donor per patient for both, the primary FMT and a scheduled booster FMT. Donors will be divided into those, who successfully improved PFS and/or tumor response versus those, who were not able to induce treatment response. Donor stool will be evaluated by 16s-RNA analysis.
Detection of specific patients' microbiota pre and post FMT leading to response. | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  Patients will be divided into responders and nonresponders and microbiota will be analyzed via 16s-RNA analysis before and after FMT. We will look into specific donor-signaling in patients stool samples after FMT, as well as trying to identify groups of intestinal microbiota associated with higher response rates to CI re-challenge.
Frequency of Adverse Events categorized according to the CTCAE grading system Version 4.0 | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  To evaluate safety and toxicity of CI therapy after FMT vs. control group. Drug toxicity will be monitored, categorized according to the CTCAE grading system Version 4.0 and managed according to recent recommendations by the SITC Toxicity Management Working Group.
Serum Neutrophil-to-Lymphocyte Ratio (NLR) pre- and post-FMT as an indicator for response. | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  In our study we will look at potential alterations in NLR after FMT and whether this can indicate response to CI treatment after FMT.
Detection of differences between primary and secondary non-responders to CI therapy and their specific outcome after FMT by performing a subgroup analysis. | 3 months after checkpoint inhibitor (CI) therapy following FMT.
  To date and according to present data we do not know, whether primary or secondary non-responders may have a better potential to respond to FMT in order to reach PFS under CI rechallenge. Hence, a subgroup analysis will be performed, in order to identify patient groups best suited for such treatment in the future.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria